CLINICAL TRIAL: NCT03902015
Title: Technology Efficacy of "Nuance Hearing" Among Students Suffering From Attention Disorders- A Pilot Study
Brief Title: "Nuance Hearing" for Attention Deficit Hyperactivity Disorder
Acronym: ADHD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Nuance Hearing (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NuanceADHD pilot
Record Dates: First submitted 2019-03-27; First posted 2019-04-03 (Actual); Last update posted 2019-04-03 (Actual); Status verified 2019-04

CONDITIONS: Attention Deficit Hyperactivity Disorder
Keywords: Attention Deficit/Hyperactivity Disorder
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Nuance Phone case (Experimental): "Nuance Hearing" has developed a technology enabling focused hearing. The Selective Noise Cancellation (SNC) technology consists of an advanced beam-forming algorithm that tones down the ambient sound by up to 15 decibels (dB) in order to focus on a primary audio source. The device consists of a special phone case(for iPhone) containing microphone array. Controlling the direction of focus is enabled through the use of a designated app. The user can place the phone case on his/hers table and can choose the direction of preferred listening, without having to ask the talker to hold the device.
  Interventions: Device: Nuance Phone case

INTERVENTIONS:
Device: Nuance Phone case — participants will receive a phone (iPhone) with the Nuance Phone case and a designated app required for the use of the device. Participants will first undergo hearing test via the app, and afterwards (in case they are not excluded based on hearing status), will receive a introduction on how to use the app and the device. Before starting the clinical trial, children will undergo three adjustments days in which they will practice using the device in school. During this period the researchers will make sure that the participants are adapting to the use of the device, and in any case there is a problem, will be able to contact a representative of "Nuance Hearing" who will be available to support technical issues.

SUMMARY:
The aim of the current study is to examine whether the ability to avoid irrelevant auditory stimuli and focus hearing, enabled by the device developed by "Nuance Hearing", may help students with ADHD in classroom listening situations by significantly reducing background distractions.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of attention deficit hyperactivity disorder (ADHD) according to Diagnostic and Statistical Manual of Mental Disorders, 5th Edition (DSM IV)
* Have fulfilled the "Test of variables of attention"
* with normal hearing

Exclusion Criteria:

* Moderate to severe co-morbid psychiatric disorders
* Neurological chronic disease

Ages: 14 Years to 17 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2019-05 (Estimated); Primary Completion 2020-01 (Estimated); Study Completion 2020-02 (Estimated)

PRIMARY OUTCOMES:
Listening inventory for education - revised (L.I.F.E - R) 1 week after baseline | 1 week after baseline
  A self-assessment questionnaire for school aged children. This version of the questionnaire was developed to assess effectiveness of sound enhancement devices in the school and other social activities. The questionnaire is comprised of 10 items (for example - how well could you hear the words the teacher is saying when there is noise from the hallway") rated in a scale of 0 to 10, where 10 - always easy and 0- always difficult.

CONTACTS AND LOCATIONS:
Overall Officials: Iris Manor, phd, Principal Investigator — Geha Mental Health Center